CLINICAL TRIAL: NCT02636738
Title: A Prospective, Multicenter, Single-arm, Non-controlled Study to Evaluate The Safety and Utility of VelaTM XL Thulium Laser in Cutting And Hemostasis For Gastrointestinal Epithelial Neoplasia In Chinese Population
Brief Title: Vela China Study: in Cutting And Hemostasis For Gastrointestinal Epithelial Neoplasia In Chinese Population
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: strategy change
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7110
Record Dates: First submitted 2015-12-11; First posted 2015-12-22 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2015-09

CONDITIONS: Indication for Modification of Patient Physical Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- experiment (Experimental): Vela XL thulium laser, laser fiber and accessories
  Interventions: Device: Vela XL thulium laser, laser fiber and accessories.

INTERVENTIONS:
Device: Vela XL thulium laser, laser fiber and accessories. — The VelaTM XL Laser is a continuous wave thulium laser that uses an optimized 1.94μm wavelength. This powerful, highly precise laser is designed for hemostatic cutting or ablation of soft and hard tissue

SUMMARY:
Prospective, multicenter, single-arm, non-controlled, 60 subjects enrolled and 14 days follow up for evaluate the safety and utility of VelaTM XL thulium laser.

DETAILED DESCRIPTION:
This study aimed to evaluate the safety and utility of VelaTM XL thulium laser in cutting and hemostasis for gastrointestinal epithelial neoplasia in Chinese population.

Vela China study will enroll at least 60 patients. Follow up points are 72 ±3 hours post procedure, 7±2 days post procedure, 14 days(±2 days) post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent to participate in the study and comply with the study procedures.
* Diagnosed as gastrointestinal epithelial neoplasia and admitted to hospital for gastrointestinal ESD procedure.
* EUS and/or CT are performed to confirm the absence of regional lymph node or distant metastasis.

Exclusion Criteria:

* Endoscopic techniques or treatment are contraindicated.
* Requirement for anticoagulation that cannot be safely stopped at least 7 days prior to the procedure.
* Based on doctor's evaluation, the patient's medical condition doesn't fit for this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Technique success | 1 hour
  The procedure is mostly completed solely at one ESD procedure by VelaTM XL thulium laser, only if the direction of the laser could not be adjacent to the target, endoscopy knives will be assisted. The technique success rate will be calculated by the ratio of operation success subjects to total enrolled subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Shutian Zhang, Principal Investigator — Beijing Friendship Hospital
Locations (2):
- China (2):
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Nanfang Hospital, Guangzhou, Guangdong